CLINICAL TRIAL: NCT07079982
Title: Effects of Freeze-dried Grape Powder on Immune Profiles in Healthy Aging Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Responsible Party: Principal Investigator, Catherine Andersen, Associate Professor, University of Connecticut
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B2024-0072/24-02-508-910
Record Dates: First submitted 2025-07-11; First posted 2025-07-23 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Healthy Aging; Inflammation
Keywords: Grapes; Healthy aging; Inflammation; Immune profiles
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Freeze-dried whole grape powder (Experimental)
  Interventions: Other: Freeze-dried whole grape powder
- Control grape-free powder (Placebo Comparator)
  Interventions: Other: Control grape-free powder

INTERVENTIONS:
Other: Freeze-dried whole grape powder — Studying the effects of freeze-dried whole grape powder on immune profiles in healthy aging adults
  Arms: Freeze-dried whole grape powder
Other: Control grape-free powder — Studying effects of a control grape-free powder on immune profiles in healthy aging
  Arms: Control grape-free powder

SUMMARY:
The purpose of this study is to investigate the effects of consuming grape powder on immune profiles in healthy middle- and older-aged individuals. Specifically, the investigators are interested in evaluating the potential effects of grapes in influencing markers of immune function, inflammation, and metabolism that are known to change with aging. Grapes contain several nutrients and antioxidant polyphenols such as resveratrol, quercetin, vitamin K and fiber, which are known to promote heart and immune health. However, the effects of grapes on altering immune profiles within the context of aging is not well understood. Therefore, this study will explore how daily grape consumption impacts certain markers of immunity in healthy middle- and older-aged adults.

The main study procedures include consumption of a freeze-dried grape powder and control powder (which tastes the same but has none of the grape compounds that are being studied) mixed with water as a beverage on a daily basis for 4 weeks each. The investigators will additionally ask that participants avoid eating grapes and certain other antioxidant/grape-related foods and beverages throughout the 13-week study. Participants will additionally be asked to complete surveys about their diet, physical activity, and medical history, as well as provide blood samples and body weight measures throughout the course of the study. Participation in the study is expected to last about 6.25 hours over the course of 13 weeks and will include 7 visits.

ELIGIBILITY:
Inclusion Criteria:

* 50-75 years old (at time of screening)
* Body mass index (BMI) 18.5 to < 30 kg/m2
* Willing to consume grape and control powder during study periods, and refrain from eating grapes and certain other polyphenol-rich foods and beverages during the study
* Do not fit any exclusion criteria

Exclusion Criteria:

* <50 years old and >75 years old
* BMI <18.5 and ≥ 30 kg/m2 or body weight < 110 pounds
* Experienced >10% weight change in the past 4 weeks
* Elevated fasting glucose levels (fasting glucose higher than 126 mg/dL) and triglycerides greater than 500 mg/dL
* Self-reported and/or physician-diagnosed history of diabetes mellitus, coronary heart disease, stroke, renal or liver disease, cancer, eating disorders, certain severe and/or relapsing/remitting autoimmune, inflammatory, or metabolic diseases, chronic infections, scleroderma, blood clotting disorders, intravenous drug use, or current pregnancy or lactation
* Allergy to grapes or any ingredients in the grape or control powders
* Implanted medical device (e.g., pacemaker) or other health condition that would prevent measurement of body composition by bioelectrical impedance
* Currently taking lipid-lowering medications (e.g., statins, fibrates), glucose-regulating medications, anti-inflammatory medications (e.g., non-steroidal anti-inflammatory drugs (NSAIDs), corticosteroids), or medications that primarily affect blood clotting (e.g., warfarin), long-term antibiotics in the last 3 months, active use of probiotics during the intervention
* Active smoker

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Concentration of lipopolysaccharide (LPS)-induced interleukin-1 beta (IL-1beta) secreted from subject-derived primary immune cells ex vivo | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nutritional Sciences, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No